CLINICAL TRIAL: NCT01563900
Title: Continuous Positive Airway Pressure for Fatigue Treatment in Patients With Multiple Sclerosis and Obstructive Sleep Apnea
Brief Title: Continuous Positive Airway Pressure (CPAP) for Fatigue in Patients With Multiple Sclerosis (MS) and Obstructive Sleep Apnea (OSA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Was unable to recruit subjects
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dr. Hryar Attarian, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00052358
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Fatigue; Multiple Sclerosis; Sleep Apnea
Keywords: fatigue; multiple sclerosis; sleep apnea; CPAP
MeSH Terms: conditions — Fatigue; Multiple Sclerosis; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham-CPAP group (Sham Comparator): The sham-CPAP device will be set at 4 centimeters of water pressure (cwp).
  Interventions: Device: Sham-CPAP
- Auto-titration CPAP (Active Comparator): This group will received an auto-titration CPAP, which will have a pressure range of 5 to 15 cwp. This device delivers pressure as needed by the patient at any given time while using the device.
  Interventions: Device: Auto-titration CPAP

INTERVENTIONS:
Device: Auto-titration CPAP — An auto-titration CPAP will be set at a pressure between 5 to 15 cwp. This device delivers pressure as needed by the patient at any given time while using the device.
  Other Names: Respironics CPAP device will be used.
  Arms: Auto-titration CPAP
Device: Sham-CPAP — The sham-CPAP device will be set at 4 centimeters of water pressure (cwp). An exhalation connector will be place between the mask interface and the tubing without the enlarged port to maintain blinding; the final pressure delivered to the participant will be 2 cwp.
  Other Names: Respironics CPAP device
  Arms: sham-CPAP group

SUMMARY:
Fatigue is a symptom present in 76 to 92% of people with multiple sclerosis (MS). Fatigue is usually described as an overwhelming sense of tiredness, lack of energy, and feeling of exhaustion which is different from sleepiness. Fatigue is also a symptom commonly seen in people with obstructive sleep apnea (OSA). The overall objective is to develop a non-pharmacological treatment for fatigue in MS. The objective of this study is to evaluate if treatment of OSA with continuous positive airway pressure (CPAP) improves fatigue in MS subjects with OSA and fatigue. This will be a small pilot randomized, double-blind, sham-controlled clinical trial; the control group will be treated with a sham-CPAP machine and intervention group will be treated with an auto-titration CPAP machine. The primary outcome measure will be improvement (decrease) in the Modified Fatigue Impact Scale from baseline. The duration of intervention will be 12 weeks to achieve a clinical response in the treatment group. After this intervention participants in both groups will be offered a referral to the sleep clinic of their preference for formal treatment as per standard of care.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a demyelinating inflammatory disease that is one of the most common neurological causes of disability in young adults. Besides physical disability, fatigue is a very common symptom present in 76 to 92% of people with MS. The 1998 Multiple Sclerosis Council for clinical practice guidelines published a consensus definition: subjective lack of physical and/or mental energy that is perceived by the individual or caregiver to interfere with the usual and desired activity. Although fatigue may be difficult to differentiate from sleepiness, it is a clinically different symptom. Sleepiness is the tendency to fall asleep or doze off. Some reports that the prevalence of moderate to severe sleep problems in MS is significantly higher than in the general population 51.5% vs 33.1%. It has also been reported that poor sleep can correlate with depression in subject with MS. Few studies have examined the effect of stimulants, amantadine or modafinil for treatment of fatigue and have shown contradictory data as effective treatments in MS patients.

Obstructive sleep apnea (OSA) has also been seen described in MS. Few case reports studies have reported that MS patients with OSA treated with continuous positive airway pressure (CPAP) had improvement in fatigue but not quality of life. Although the prevalence of OSA in the MS population is unknown, it may as much as twice as common as in the general population, which is 3 to 7%. Aside from the increased risk of daytime sleepiness, mood disorders, cardiovascular risk factors and accidents, OSA has also been implicated in increasing inflammatory markers like tumor necrosis factor (TNF-α). Elevation in TNF-α has also been seen in MS patients complaining of fatigue, which is thought to play a role in pathophysiology of fatigue in MS. The rational of this study is to determine if treatment of OSA with CPAP in MS patients improves fatigue. If effective, CPAP may not only decrease the risk of long term complications but may also improve the quality of life and daily living of these patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Diagnosis of clinical MS as defined by the 2010 McDonald criteria
* Have either relapsing remitting, primary progressive or secondary progressive forms of MS
* expanded disability status scale ≤5
* Complaint of fatigue defined subjective lack of physical and/or mental energy that is perceived by the individual or caregiver to interfere with the usual and desired activity.
* Berlin questionnaire score of ≥2 35
* Mild to moderate OSA defined as Apnea hypopnea index (AHI) of ≥ 5 and < 30 events/hour on baseline ambulatory PSG

Exclusion Criteria:

* Prior diagnosis, past or current treatment for sleep related breathing disorder
* Severe sleep apnea defined as AHI ≥ 30 events/hour on baseline ambulatory PSG,
* Prior diagnosis of restless leg syndrome, parasomnias, insomnia, and narcolepsy
* Prior diagnosis of pulmonary disease: asthma, chronic obstructive pulmonary disease and bronchiectasis
* Diagnosis of clinical depression or Center for epidemiologic studies-depression scale(CES-D)score of ≥ 16 36,37
* An acute MS exacerbation in the last 3 months. If patient has an acute exacerbation during the study, the patient will be excluded from the study as this can be a cause fatigue
* Started on any disease modifying treatment (either primary or second line agents) or have switched to a second therapy in the last 6 month poor sleep and fatigue can be side effects.
* Current use of sedative-hypnotics medications, tricyclic, antidepressants, or trazodone.
* Started or change in dose within the last 3 months of amantadine, modafinil, armodafinil, or other stimulating agent for MS related fatigue
* Pregnancy
* Unstable medical or psychiatric condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
10 point change in Modified Fatigue Impact Scale (MFIS) | 78 ± 7 days

SECONDARY OUTCOMES:
Improvement in the Epworth sleeping scale (ESS). | 78 ± 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Hrayr Attarian, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern UNiversity, Department of Neurology, Chicago, Illinois, United States

REFERENCES:
- [Background] Krupp LB, Coyle PK, Doscher C, Miller A, Cross AH, Jandorf L, Halper J, Johnson B, Morgante L, Grimson R. Fatigue therapy in multiple sclerosis: results of a double-blind, randomized, parallel trial of amantadine, pemoline, and placebo. Neurology. 1995 Nov;45(11):1956-61. doi: 10.1212/wnl.45.11.1956. PMID 7501140
- [Background] Reder AT, Antel JP. Clinical spectrum of multiple sclerosis. Neurol Clin. 1983 Aug;1(3):573-99. PMID 6095009
- [Background] Krupp LB, Serafin DJ, Christodoulou C. Multiple sclerosis-associated fatigue. Expert Rev Neurother. 2010 Sep;10(9):1437-47. doi: 10.1586/ern.10.99. PMID 20819014
- [Background] Shahid A, Shen J, Shapiro CM. Measurements of sleepiness and fatigue. J Psychosom Res. 2010 Jul;69(1):81-9. doi: 10.1016/j.jpsychores.2010.04.001. PMID 20630266
- [Background] Attarian HP, Brown KM, Duntley SP, Carter JD, Cross AH. The relationship of sleep disturbances and fatigue in multiple sclerosis. Arch Neurol. 2004 Apr;61(4):525-8. doi: 10.1001/archneur.61.4.525. PMID 15096400
- [Background] Bamer AM, Johnson KL, Amtmann DA, Kraft GH. Beyond fatigue: Assessing variables associated with sleep problems and use of sleep medications in multiple sclerosis. Clin Epidemiol. 2010 May 1;2010(2):99-106. doi: 10.2147/CLEP.S10425. PMID 20838467
- [Background] Merlino G, Fratticci L, Lenchig C, Valente M, Cargnelutti D, Picello M, Serafini A, Dolso P, Gigli GL. Prevalence of 'poor sleep' among patients with multiple sclerosis: an independent predictor of mental and physical status. Sleep Med. 2009 Jan;10(1):26-34. doi: 10.1016/j.sleep.2007.11.004. Epub 2008 Jan 22. PMID 18207453
- [Background] Rammohan KW, Rosenberg JH, Lynn DJ, Blumenfeld AM, Pollak CP, Nagaraja HN. Efficacy and safety of modafinil (Provigil) for the treatment of fatigue in multiple sclerosis: a two centre phase 2 study. J Neurol Neurosurg Psychiatry. 2002 Feb;72(2):179-83. doi: 10.1136/jnnp.72.2.179. PMID 11796766
- [Background] Jackson ML, Stough C, Howard ME, Spong J, Downey LA, Thompson B. The contribution of fatigue and sleepiness to depression in patients attending the sleep laboratory for evaluation of obstructive sleep apnea. Sleep Breath. 2011 Sep;15(3):439-45. doi: 10.1007/s11325-010-0355-2. Epub 2010 May 6. PMID 20446116
- [Background] Kohli P, Balachandran JS, Malhotra A. Obstructive sleep apnea and the risk for cardiovascular disease. Curr Atheroscler Rep. 2011 Apr;13(2):138-46. doi: 10.1007/s11883-011-0161-8. PMID 21253882
- [Background] Tamaki S, Yamauchi M, Fukuoka A, Makinodan K, Koyama N, Tomoda K, Yoshikawa M, Kimura H. Production of inflammatory mediators by monocytes in patients with obstructive sleep apnea syndrome. Intern Med. 2009;48(15):1255-62. doi: 10.2169/internalmedicine.48.2366. Epub 2009 Aug 3. PMID 19652426
- [Background] Heesen C, Nawrath L, Reich C, Bauer N, Schulz KH, Gold SM. Fatigue in multiple sclerosis: an example of cytokine mediated sickness behaviour? J Neurol Neurosurg Psychiatry. 2006 Jan;77(1):34-9. doi: 10.1136/jnnp.2005.065805. PMID 16361589
- [Background] Kaminska M, Kimoff RJ, Benedetti A, Robinson A, Bar-Or A, Lapierre Y, Schwartzman K, Trojan DA. Obstructive sleep apnea is associated with fatigue in multiple sclerosis. Mult Scler. 2012 Aug;18(8):1159-69. doi: 10.1177/1352458511432328. Epub 2011 Dec 19. PMID 22183937